CLINICAL TRIAL: NCT06449885
Title: A Prospective, Multi-center, Cohort Study in Newly Diagnosed Marginal Zone B-cell Lymphoma
Brief Title: A Cohort Study in Newly Diagnosed MZL
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor, Fudan University
Other Study IDs: SHCA-MZL-001
Record Dates: First submitted 2024-05-30; First posted 2024-06-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue, peripheral blood samples or bone marrow samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed marginal zone lymphoma: Newly diagnosed marginal zone lymphoma，including Mucosa-associated lymphoid tissue (MALT) lymphoma, spleen MZL, and lymph node MZL, as well as primary cutaneous MZL, and pediatric NMZL.
  Interventions: Other: patients receive optimal treatment or follow-up according to the characteristics of the disease

INTERVENTIONS:
Other: patients receive optimal treatment or follow-up according to the characteristics of the disease — Patients with MZL who are eligible for enrollment will be evaluated by the investigator and the enrolled patients will receive long-term follow-up after collecting medical history information, biological samples, and oncology data according to the study protocol. This study does not specify a detailed treatment modality, and patients receive optimal treatment or follow-up according to the characteristics of the disease.

SUMMARY:
Describe the clinical features, diagnosis and treatment status, disease course and primary outcomes of different subtypes of marginal zone B-cell lymphoma (MZL), observe the therapeutic efficacy and safety of different treatment modalities.

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) originates from the marginal zone of lymphatic follicles and can occur in the spleen, lymph nodes and mucosal lymphoid tissues, and the incidence increases with age. The clinicopathological features of each subtype of MZL are heterogeneous, and their clinical manifestations, biology, etiology, and treatment are all quite heterogeneous, and there is still significant uncertainty about the optimal treatment pathway. This prospective, multicenter, cohort study aims to describe the clinical features, diagnosis and treatment status, disease course and primary outcomes of different subtypes of MZL, and to observe the therapeutic efficacy and safety of different treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years old; Male or female.
* Newly diagnosed marginal zone lymphoma by histopathology within the past 6 months (180 days) and no anti-tumor therapy (including chemotherapy, radiotherapy, and biological therapy or immunotherapy for the treatment of tumors).
* Willing to provide biological samples required for the study, including blood samples and tumor tissue.
* Voluntarily join this study and sign the informed consent form.
* Willing to accept long-term follow-up.

Exclusion Criteria:

* Patients with HIV infection.
* Those who cannot come to the hospital regularly for follow-up.
* Those with comorbidities and speech impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed marginal zone lymphoma who are eligible for enrollment will be evaluated by the investigator and the enrolled patients will receive long-term follow-up after collecting medical history information, biological samples, and oncology data according to the study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | assessed up to 10 years
  record the period from date of patients sign informed consent until the date of documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Time to treatment | assessed up to 10 years
  calculate the time interval between the start of diagnosis and the first dose of anti-tumor therapy.
Time to next treatment | assessed up to 10 years
  the time interval from initiation of treatment to initiation of next-line anti-neoplastic therapy or death due to any cause.
ORR | up to 6 months
  the ratio of numbers of patients with complete response and partial response to all the participants receiving treatment
Overall survival | assessed up to 10 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time
Adverse events | Throughout the treatment period, up to 10 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0
Histologic transformation rate | Throughout the study, up to 10 years
  Proportion of patients with histologic transformation in all patients
Occurrence rate of a second tumor | Throughout the study, up to 10 years
  Proportion of patients with a second tumor in all patients

OTHER OUTCOMES:
serum biomarkers | Throughout the study, up to 10 years
  detection of serum DNA biomarkers in the treatment of marginal zone lymphoma
tissue biomarkers | Throughout the study, up to 10 years
  detection of tissue DNA biomarkers in the treatment of marginal zone lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, M.D, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China